CLINICAL TRIAL: NCT01152814
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated, Adjuvanted With MF59C.1 Influenza Vaccine, Formulation 2010-2011, When Administered to Elderly Subjects
Brief Title: Study to Evaluate Safety and Immunogenicity of Sub-unit Adjuvanted Influenza Vaccine Administered to Elderly Subjects, Formulation 2010-2011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V70_25S; 2010-018603-29 (EudraCT Number)
Record Dates: First submitted 2010-06-28; First posted 2010-06-29 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Seasonal Influenza
Keywords: Seasonal influenza; Vaccine

ARMS (1):
- Arm 1 (Experimental): No comparator is administered, only one IM single dose of trivalent subunit inactivated influenza vaccine is administered during the vaccination visit
  Interventions: Biological: Seasonal flu vaccine

INTERVENTIONS:
Biological: Seasonal flu vaccine — This phase II is performed as a multicenters study site in elderly subjects. Enrolled subjects received one single IM dose of trivalent subunit inactivated adjuvanted flu vaccine during the vaccination visit, according to the study protocol (follow-up period: till day 22)

SUMMARY:
This study will evaluate the safety and immunogenicity of a sub-unit, adjuvanted influenza vaccine administered to elderly subjects

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females volunteers of 65 years of age or older
* Mentally competent
* Willing and able to give written informed consent prior to study entry.
* Able to comply with all the study requirements.
* In general good health

Key Exclusion Criteria:

* Any serious chronic or acute disease
* History of any anaphylactic reaction and/or serious allergic reaction following a vaccination
* Known or suspected impairment/alteration of immune function
* Bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject
* Within the past 6 months, they have had laboratory confirmed influenza disease or received influenza vaccine
* Fever (i.e., axillary temperature ≥38°C) within the last 3 days of intended study vaccination
* Individuals who received any other vaccines within 4 weeks prior to enrollment in this study or who are planning to receive any vaccine within 4 weeks from the study vaccines

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G. D'Annunzio, Via dei Vestini, Chieti
  - Dipartimento di Medicina Clinica e Sperimentale - Sezione di Igiene e Medicina Preventiva, Via Fossato di Mortara, 64/b, Ferrara
  - Dipartimento di Scienze della Salute Università di Genova Via Pastore, 1, Genova
  - Centro Satellite. ASL Lanciano - Vasto, sede legale Via S. Spaventa, 37, Lanciano
  - Centro Satellite. Distretto Sanitario di Base di Fossacesia in Via Polidoro-Vasto, Lanciano
  - Vaccine and Immunotherapy Research Center Department of Infectious and Tropical Diseases San Raffaele Scientific Institute Via Stamira d'Ancona, 20, Milan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 64 participants ≥65 years of age were enrolled at 5 sites in Italy.
Pre-assignment Details: Blood samples for the determination of antibody titers were obtained prior to vaccination.
Groups:
- FLUAD: Participants received a single intramuscular (IM) dose of 0.5 milliliter (mL) of FLUAD containing 15μg each of the three influenza antigens into the deltoid region of the non-dominant arm during the vaccination visit, according to the study protocol until Day 22.
Period: Overall Study
Arm/Group | FLUAD
Started | 64
Completed | 62
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were enrolled and randomized into the study.
Groups:
- FLUAD: Participants received a single IM dose of 0.5 mL of FLUAD containing 15μg each of the three influenza antigens into the deltoid region of the non-dominant arm during the vaccination visit, according to the study protocol until Day 22.
Arm/Group | FLUAD
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.3 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Seroconversion or Significant Increase in Single Radial Hemolysis (SRH) Area Against Each of Three Vaccine Strains After One Vaccination of FLUAD
Description: Immunogenicity was measured as the percentage of participants who achieved seroconversion or significant increase in single radial hemolysis (SRH) area, against each of the three vaccine strains, three weeks after vaccination (day 22), evaluated using SRH assay. Seroconversion: proportion of participants with negative pre-vaccination serum and a post-vaccination serum area ≥ 25 mm2. Significant increase: proportion of participants with at least a 50% increase in area from positive pre-vaccination serum. Seroconversion or significant increase: proportion of participants with either seroconversion or significant increase.
  The European (Committee for Medicinal Products for Human Use [CHMP]) criterion is met, if percentage of participants achieving seroconversion or significant increase in SRH area is 30% (≥65 years).
Time Frame: day 22
Population: Per protocol (PP) analysis set included all enrolled participants who had received the vaccine, provided evaluable serum samples before and after vaccination, and had no major protocol violation.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLUAD
Number analyzed (Participants) | 62
Percentage of participants
  A/H1N1 | 45 [32 to 58]
  A/H3N2 | 61 [48 to 73]
  B | 27 [17 to 40]

2. Secondary Outcome: Number of Participants Who Reported Solicited Local and Systemic Reactions
Description: Safety was assessed for all participants who reported solicited local and systemic reactions from Day 1 up to and including Day 4 after the FLUAD vaccination in accordance with available safety data on influenza vaccines.
Time Frame: 1 to 4 days post-vaccination
Population: Analysis was done using the safety dataset; all participants exposed and who had post-baseline safety data were included in the safety analysis.
Measure: Number; unit: Number of participants
Arm/Group | FLUAD
Number analyzed (Participants) | 64
Number of participants
  Injection site ecchymosis (N= 62) | 2
  Injection site erythema (N= 62) | 4
  Injection site induration (N= 62) | 2
  Injection site swelling (N= 62) | 0
  Injection site pain (N= 62) | 15
  Chills/Shivering (N= 62) | 2
  Malaise (N= 62) | 2
  Myalgia (N= 62) | 7
  Arthralgia (N= 62) | 4
  Headache (N= 62) | 5
  Sweating (N= 62) | 7
  Fatigue (N= 62) | 5
  Fever (≥38°C) (N= 59) | 0

3. Primary Outcome: Geometric Mean Ratio of Participants Against Each of the Three Vaccine Strains After One Vaccination of FLUAD
Description: Geometric mean ratio (GMR) of participants was calculated as the ratio of post-vaccination to pre-vaccination SRH geometric mean areas (GMAs), directed against each of the three vaccine strains, three weeks after FLUAD vaccination (day 22).
  The CHMP criterion was met if the geometric mean increase (GMR, day 22/day 1) in SRH antibody area is >2.0 (≥65 years).
Time Frame: day 22
Population: Analysis was done using the PP dataset.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | FLUAD
Number analyzed (Participants) | 62
Ratio
  A/H1N1 | 1.96 [1.59 to 2.42]
  A/H3N2 | 1.88 [1.64 to 2.16]
  B | 1.32 [1.22 to 1.43]

4. Primary Outcome: Percentage of Participants Who Achieved SRH Area ≥25mm2 Against Each of the Three Vaccine Strains After One Vaccination of FLUAD
Description: Immunogenicity was measured as the percentage of participants achieving SRH area ≥25 mm2 against each of the three vaccine strains at baseline (day 1) and three weeks after FLUAD vaccination (day 22).
  This criterion is met according to CHMP guideline if percentage of participants achieving SRH area ≥25 mm2 is 60% (≥65 years).
Time Frame: day 22
Population: Analysis was done using the PP dataset.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FLUAD
Number analyzed (Participants) | 62
Percentage of participants
  A/H1N1 | 97 [89 to 100]
  A/H3N2 | 71 [58 to 82]
  B | 100 [94 to 100]

ADVERSE EVENTS:
Time Frame: From Day 1 through Day 22.
Description: Adverse events other than local and systemic reactions or solicited reactions lasting longer than 4 days after vaccination were documented during the study period. Analysis was done using the safety dataset; all participants exposed and who had post-baseline safety data were included in the safety analysis.
Arm/Group | FLUAD
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 4/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLUAD (N=64)
Fatigue (General disorders) | 2
Malaise (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.